CLINICAL TRIAL: NCT06492759
Title: A Phase II Study of High Dose Radiotherapy in Combination With Pembrolizumab Plus Chemotherapy in Patients With PD-L1 Positive Metastatic Triple Negative Breast Cancer
Brief Title: High Dose Radiation Therapy With Pembrolizumab and Chemotherapy for the Treatment of Patients With PD-L1 Positive Metastatic Triple Negative Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Manali Bhave, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005578; P30CA138292 (NIH); WINSHIP5835-22 (Other: Emory University Hospital/Winship Cancer Institute)
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-10

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Radiotherapy; Radiation; Therapeutics; pembrolizumab; Immunoglobulin G; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes; Paclitaxel; Carboplatin; Gemcitabine; Biopsy; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (radiation, pembrolizumab, chemotherapy) (Experimental): Patients undergo radiation therapy once every other day for 3 doses. Beginning within 48 hours of their first dose of radiation therapy, patients receive standard of care pembrolizumab IV on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also receive 1 of 3 standard of care chemotherapy options: nab-paclitaxel IV on days 1, 8, and 15 of each cycle, or paclitaxel IV on days 1, 8, and 15 of each cycle, or carboplatin IV and gemcitabine IV on days 1 and 8 of each cycle. Cycles of nab-paclitaxel and paclitaxel repeat every 28 days and cycles of carboplatin and gemcitabine repeat every 21 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo a biopsy at baseline and 2 weeks after radiation therapy and also undergo CT scans, bone scans and blood sample collections throughout the trial.
  Interventions: Radiation: Radiation Therapy; Biological: Pembrolizumab; Drug: Nab-paclitaxel; Drug: Paclitaxel; Drug: Carboplatin; Drug: Gemcitabine; Procedure: Biopsy; Procedure: Computed Tomography; Procedure: Bone Scan; Procedure: Biospecimen Collection; Other: Medical Chart Review

INTERVENTIONS:
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy, Energy Type, Irradiate, Irradiated, irradiation, Radiation, Radiation Therapy, Therapy, Radiotherapeutics, Radiotherapy, RT, Therapy, Radiation
Biological: Pembrolizumab — Given IV
  Other Names: 1374853-91-4, BCD-201, Immunoglobulin G4, Anti-(Human Programmed Cell Death 1); Humanized Mouse Monoclonal (228-L-proline(H10-S>P))gamma 4 Heavy Chain (134-218')-disulfide with Humanized; Monoclonal Kappa Light Chain Dimer (226-226'':229-229'')-bisdisulfide, Keytruda, Lambrolizumab, MK-3475, PEMBROLIZUMAB, Pembrolizumab, Biosimilar BCD-201, SCH 900475
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007, ABI-007, ABI-007, Abraxane, Abraxane, Albumin-bound Paclitaxel, Albumin-Stabilized Nanoparticle Paclitaxel, Nanoparticle Albumin-bound; Paclitaxel, nanoparticle paclitaxel, Nanoparticle Paclitaxel, Paclitaxel Albumin, paclitaxel albumin-stabilized nanoparticle formulation, Paclitaxel nanoparticle albumin-bound,; Paclitaxel Protein-Bound, protein-bound paclitaxel, Protein-bound Paclitaxel
Drug: Paclitaxel — Given IV
  Other Names: 33069-62-4,5Beta,20-epoxy-1,2alpha,4,7beta,10beta,13alpha-hexahydroxytax-11-en-9-one,4,10-Diacetate 2-Benzoate 13-Ester with (2R,3S)-N-Benzoyl-3-phenylisoserine, [2aR-[2a Alpha,4beta,4a beta,6beta
Drug: Carboplatin — Given IV
  Other Names: SP-4-2)-diammine[1,1-cyclobutanedicarboxylato(2--)-O,O']platinum, 1,1-cyclobutanedicarboxylic acid platinum complex, 41575-94-4, Blastocarb, Carboplat, CARBOPLATIN,; Hexal, Carboplatino, Carboplatinum, Carbosin, Carbosol, Carbotec, CBDCA, CBDCA, cis-diammine(1,1-cyclobutanedicarboxylato) platinum(II),; complex, 41575-94-4, Blastocarb, Carboplat, CARBOPLATIN, Carboplatin, Carboplatin Hexal, Carboplatino, Carboplatinum,; Carbosin, Carbosol, Carbotec, CBDCA, cis-diammine(1,1-cyclobutanedicarboxylato) platinum(II), Cis-Diammine(cyclobutane-1,1-dicarboxylato)platinum,
Drug: Gemcitabine — Given IV
  Other Names: 1-(2-Oxo-4-amino-1,2-dihydropyrimidin-1-yl)-2-deoxy-2,2-difluororibose, 2'Deoxy-2',2'-Difluorocytidine, 95058-81-4, dFdC, dFdCyd, Difluorodeoxycytidine, Gemcitabine, GEMCITABINE,
Procedure: Biopsy — Undergo biopsy
  Other Names: Biopsy, BIOPSY_TYPE
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT, CAT Scan, Computed Axial Tomography, Computed Tomography, Computerized Axial Tomography,Computerized Axial Tomography,
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scan, bone scan, Bone Scan, Bone Scan, Bone Scan, Bone Scintigraphy
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection, Biological Sample Collection, Biospecimen Collected, Biospecimen Collection, Specimen Collection
Other: Medical Chart Review — Ancillary studies
  Other Names: Chart Review, Medical Chart Review

SUMMARY:
This phase II trial tests how well radiation therapy with pembrolizumab and chemotherapy (paclitaxel or nab-paclitaxel or carboplatin and gemcitabine) works in treating patients with PD-L1 positive triple negative breast cancer that has spread from where it first started (primary site) to other places in the body (metastatic). Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill tumor cells and shrink tumors. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the tumor, and may interfere with the ability of tumor cells to grow and spread. Paclitaxel is in a class of medications called antimicrotubule agents. It stops cancer cells from growing and dividing and may kill them. Nab-paclitaxel is an albumin-stabilized nanoparticle formulation of paclitaxel which may have fewer side effects and work better than other forms of paclitaxel. Carboplatin is in a class of medications known as platinum-containing compounds. It works by killing, stopping or slowing the growth of cancer cells. Gemcitabine is a chemotherapy drug that blocks the cells from making DNA and may kill cancer cells. High dose radiation therapy with pembrolizumab and chemotherapy may effective in treating patients with PD-L1 positive metastatic triple negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the 12 month progression-free survival (PFS) in PD-L1 positive, triple negative breast cancer patients treated with high dose radiotherapy before and concurrently with the first cycle of pembrolizumab plus chemotherapy.

SECONDARY OBJECTIVES:

I. To evaluate the objective response rate (ORR) in non-irradiated lesions nine weeks after the first dose of pembrolizumab in PD-L1 positive, triple negative breast cancer patients treated with high dose radiotherapy before and concurrently with the first cycle pembrolizumab plus chemotherapy (ORR per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1).

II. To determine if targeted, high dose radiotherapy to up to 3 metastatic sites in combination with pembrolizumab plus chemotherapy in patients with metastatic triple negative breast cancer (> 2 sites) adversely increases the frequency and severity of toxicities associated with radiotherapy or pembrolizumab plus chemotherapy when administered separately.

III. To determine progression-free survival (PFS) in breast cancer patients treated with high dose radiotherapy, pembrolizumab, and chemotherapy.

EXPLORATORY OBJECTIVES:

I. To collect, store, and analyze circulating tumor deoxyribonucleic acid (ctDNA) in metastatic breast cancer patients treated with radiotherapy, pembrolizumab, and chemotherapy to determine the relationship between ctDNA and PFS and ORR.

II. To collect, store and analyze tumor tissue from a non-irradiated metastatic breast cancer site before and after radiotherapy to explore the immune tumor microenvironment and the immunoscore, and the relationship between the immunoscore and ORR and PFS in metastatic breast cancer patients treated with pembrolizumab and chemotherapy.

OUTLINE:

Patients undergo radiation therapy once every other day for 3 doses. Beginning within 48 hours of their first dose of radiation therapy, patients receive standard of care pembrolizumab intravenously (IV) on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also receive 1 of 3 standard of care chemotherapy options: nab-paclitaxel IV on days 1, 8, and 15 of each cycle, or paclitaxel IV on days 1, 8, and 15 of each cycle, or carboplatin IV and gemcitabine IV on days 1 and 8 of each cycle. Cycles of nab-paclitaxel and paclitaxel repeat every 28 days and cycles of carboplatin and gemcitabine repeat every 21 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo a biopsy at baseline and 2 weeks after radiation therapy and also undergo computed tomography (CT) scans, bone scans and blood sample collections throughout the trial.

After completion of study treatment, patients are followed up every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven metastatic PD-L1 positive triple negative breast cancer with at least 2 sites of measurable metastatic disease on imaging

  * Estrogen receptor (ER) and progesterone receptor (PR) negativity are defined as ≤ 10% of cells expressing hormonal receptors via immunohistochemistry (IHC) analysis
  * HER2 negativity is defined as either of the following by local laboratory assessment

    * In situ hybridization (ISH) non-amplified (ratio of HER2 to CEP17 < 2.0 or single probe average HER2 gene copy number < 4 signals/cell) or
    * IHC 0 or IHC 1+. If more than one test result is available and not all results meet the inclusion criterion definition, all results should be discussed with the Medical Monitor to establish eligibility of the patient
* PD-L1 positive as defined by Dako 22c3 assay PD-L1 combined positive score (CPS) ≥ 10
* Appropriate stage for study entry based on the following diagnostic workup:

  * History and physical examination within 60 days prior to registration
  * Clinical grade CT scans of the chest, abdomen, and pelvis with radionuclide bone scan or whole body positron emission tomography (PET)/CT documenting metastatic disease within 4 weeks of the start of radiotherapy on this protocol with or without magnetic resonance imaging (MRI), as needed, documenting site of metastatic disease to be treated on protocol
* Patient must be eligible for radiotherapy as determined by their treating physician
* Patient must be eligible for immunotherapy and taxane chemotherapy as determined by their treating physician
* At least 1 metastatic site amenable to high dose radiotherapy
* Be willing and able to provide written informed consent for the trial
* Ages ≥ 18 years of age
* Biopsy proven metastatic PD-L1 positive triple negative breast cancer with at least 2 sites of measurable metastatic disease on imaging

  * Estrogen receptor (ER) and progesterone receptor (PR) negativity are defined as ≤ 10% of cells expressing hormonal receptors via immunohistochemistry (IHC) analysis
  * HER2 negativity is defined as either of the following by local laboratory assessment

    * In situ hybridization (ISH) non-amplified (ratio of HER2 to CEP17 < 2.0 or single probe average HER2 gene copy number < 4 signals/cell) or
    * IHC 0 or IHC 1+. If more than one test result is available and not all results meet the inclusion criterion definition, all results should be discussed with the Medical Monitor to establish eligibility of the patient
* PD-L1 positive as defined by Dako 22c3 assay PD-L1 combined positive score (CPS) ≥ 10
* Appropriate stage for study entry based on the following diagnostic workup:

  * History and physical examination within 60 days prior to registration
  * Clinical grade CT scans of the chest, abdomen, and pelvis with radionuclide bone scan or whole body positron emission tomography (PET)/CT documenting metastatic disease within 4 weeks of the start of radiotherapy on this protocol with or without magnetic resonance imaging (MRI), as needed, documenting site of metastatic disease to be treated on protocol
* Patient must be eligible for radiotherapy as determined by their treating physician
* Patient must be eligible for immunotherapy and taxane chemotherapy as determined by their treating physician
* At least 1 metastatic site amenable to high dose radiotherapy
* Be willing and able to provide written informed consent for the trial
* Ages ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-2, Karnofsky performance status (KPS) ≥ 60%
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST, version 1.1)
* Absolute neutrophil count ≥ 1500/mcL (obtained within 14 days prior to first study treatment)
* Platelet count ≥ 100,000/mcL (obtained within 14 days prior to first study treatment)
* Hemoglobin ≥ 9.0 g/dL (obtained within 14 days prior to first study treatment) (Note: The use of transfusion or other intervention to achieve hemoglobin [Hgb] ≥ 9.0g/dL is acceptable)
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 x the upper limit of normal (ULN) with the following exceptions (obtained within 14 days prior to first study treatment):

  * Patients with documented liver metastases: AST and ALT ≤ 5 x ULN
* Serum bilirubin ≤ 1.5 x ULN (obtained within 14 days prior to first study treatment)

  * Patients with known Gilbert disease who have serum bilirubin level ≤ 3 x ULN may be enrolled
* Calculated creatinine clearance ≥ 30 mL/min (obtained within 14 days prior to first study treatment)
* For females of child-bearing potential, negative serum or urine pregnancy test within 14 days prior to radiation simulation
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry
* Prior Treatment:

  * Patients may or may not have received radiotherapy or neoadjuvant or adjuvant chemotherapy in the treatment of their initial, non-metastatic breast cancer, but must be entered on study after their last dose of radiotherapy, last cycle of chemotherapy and biologic therapy (if applicable) and have sufficient resolution of side effects per physician assessment at time of radiotherapy. Prior immunotherapy for treatment of early stage breast cancer is allowed if metastatic recurrence occurs ≥ 6 months after last dose of immunotherapy
  * Patients must have not active wound healing issues from surgery and sufficient resolution of surgical side effects, per physician assessment, at time of radiotherapy
  * Patients are not eligible if they have received chemotherapy in the advanced/metastatic setting
  * During radiotherapy, no other investigation or commercial agents or therapy for cancer other than bisphosphonate or receptor activator nuclear kappaB ligand (RANK-L) inhibitor, pembrolizumab, and nab-paclitaxel, paclitaxel, carboplatin or gemcitabine should be administered
  * Patients may have received bisphosphonates or rank ligand inhibitors prior to enrollment on study

Exclusion Criteria:

* Prior chemotherapy or targeted therapy for metastatic triple negative breast cancer before start of pembrolizumab plus partner chemotherapy. Prior chemotherapy (including taxanes) administered in the context of curative therapy (if treatment was completed > 6 months) prior to enrollment into the trial is allowed
* Previous radiation to the metastases to be treated with radiation on this protocol
* Untreated central nervous system (CNS) disease (patients with stable CNS disease for at least 28 days and asymptomatic treated CNS metastases are permitted)
* Uncontrolled pleural effusion, pericardial effusion or ascites

  * Patients with indwelling catheters (e.g., Pleurx) are allowed
* Uncontrolled hypercalcemia (> 1.5 mmol/L ionized calcium or calcium > 12 mg/dL or corrected serum calcium > ULN) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab

  * Patients who are receiving bisphosphonate therapy specifically to prevent skeletal prevents and who do not have a history of clinically significant hypercalcemia are eligible
* History (Hx) of autoimmune disease that has required systemic treatment (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g.., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Use of chronic systemic glucocorticoid or immunosuppressive medications at time of enrollment (prednisone or equivalent steroid dose of > 10mg for > 2 weeks)
* Prior allogeneic stem cell or solid organ transplantation
* Severe, active co-morbidity such as congestive heart failure (CHF) or unstable angina within last 6 months, transmural myocardial infarction (MI) within the last 6 months
* Acute bacterial or fungal infection requiring IV antibiotics at time of registration
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan

  * History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Chronic obstructive pulmonary disease (COPD) or other respiratory illness requiring hospitalization at time of registration
* HIV positive with CD4 count < 200 cells/ microliter
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy. Indolent cancers (such as low risk prostate or in-situ cancers) that are not being treated, are acceptable
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator. Examples include:

  * Major surgical procedure within 28 days prior to randomization or anticipation of the need for a major surgical procedure during the course of the study other than for diagnosis
  * Known hypersensitivity to nab-paclitaxel or to any of the excipients
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 90 days after the last dose of trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-02-12 (Estimated); Study Completion 2028-02-13 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From start of radiation therapy to progression or death, assessed at 1 year
  Progressive disease will be determined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1. PFS will be estimated using the Kaplan-Meier method, and a 95% confidence interval for 1-year PFS will be estimated using the Greenwood formula. The 1-year PFS estimate will be compared to a null value of 30% using a one-sample log-rank test.

SECONDARY OUTCOMES:
Objective response rate (ORR) | At 9 weeks after first dose of pembrolizumab
  Response will be defined by partial or complete response on imaging using RECIST version 1.1. ORR will be estimated as a proportion, with an exact 95% confidence interval estimated using the Clopper-Pearson method.
Overall survival (OS) | From start of radiation therapy to death, assessed up to 2 years
  OS will be estimated using the Kaplan-Meier method, and median survival will be calculated. A 95% confidence interval will be estimated using the Brookmeyer-Crowley approach.
Incidence of adverse events (AEs) | Up to 90 days after the last dose of study treatment
  AEs will be determined according to the National Cancer Institute Common Terminology Criteria for Adverse Events v5. Frequencies and percentages will be used to summarize safety events.

CONTACTS AND LOCATIONS:
Overall Officials: Manali Bhave, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States